CLINICAL TRIAL: NCT05559489
Title: Implementation of an Enteral Resuscitation Bundle for the Moderate-sized Burn at Kirtipur Hospital, Nepal
Brief Title: Enteral Resuscitation Nepal
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Raslina Shreshtha, Global Health Research Fellow, Nepal Health Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010934-A
Record Dates: First submitted 2022-09-19; First posted 2022-09-29 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Burn Body Region Unspecified; Burn Shock
Keywords: Burns; Enteral Resuscitation; Oral Rehydration Solution; Burn Shock; Austere condition; Low and middle income countries
MeSH Terms: conditions — Burns; Osteoarthritis | interventions — World Health Organization oral rehydration solution; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: hybrid type 1 effectiveness-implementation study of a randomized trial of enteral-based resuscitation (intervention arm) vs. IV fluid resuscitation (standard-of-care arm) for moderate-sized burn injuries.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enteral-based Protocolized Resuscitation (Experimental): Administration of Enteral-based Resuscitation using Oral Rehydration Solution (ORS) either by mouth or via naso-enteric access for moderate sized burn injuries (15-40% TBSA) per resuscitation protocol for burn-injured patients. Resuscitation will be administered in the acute resuscitation phase of burn injury (24-72 hours post injury). Patients will receive supplemental Intravenous Fluid (IV Fluid) resuscitation using Lactated Ringer's solution as needed per protocol.
  Interventions: Drug: Oral Rehydration Solution; Drug: Lactated Ringer
- Intravenous Fluid Protocolized Resuscitation (Active Comparator): Administration of Intravenous Fluid using Lactated Ringer's solution per standard of care resuscitation protocol for patients with moderate sized burn injuries (15-40% TBSA).
  Interventions: Drug: Lactated Ringer

INTERVENTIONS:
Drug: Oral Rehydration Solution — Effectiveness- implementation study of Enteral-based resuscitation with Oral Rehydration Solution (ORS) vs standard-of-care Intravenous Fluid resuscitation for moderate-sized burn injuries in Nepal
  Other Names: Enteral-based Resuscitation
  Arms: Enteral-based Protocolized Resuscitation
Drug: Lactated Ringer — Standard-of-care Intravenous Fluid resuscitation
  Other Names: Intravenous Fluid Resuscitation

SUMMARY:
Nepal and the South Asian sub-continent carry some of the highest rates of burn injury globally, with associated high morbidity and mortality. Nepal currently has one major center equipped for comprehensive burn care, in Kirtipur, Nepal, and receives patients who are referred from around the country. At the time of presentation, most patients with major burns have had minimal to no resuscitation on arrival, and often present hours to days after the burn injury was sustained. Timely fluid resuscitation, initiated as soon as possible after a major burn injury, is the main tenet of acute burn care. Lack of adequate resuscitation in major burn injuries leads to kidney injury, progression of burn injury, sepsis, burn shock, and death. The current standard of care for major burn resuscitation is intravenous fluid resuscitation. However, in low- and middle-income countries such as Nepal, adequately trained and equipped hospitals for the treatment of burn care are not widely available (for a variety of reasons). Additionally, there is no systematic emergency medical transport system available to provide medical care and resuscitation during transport. Enteral-based resuscitation-drinking or administering fluids via the gastrointestinal tract-with substances like the WHO Oral Rehydration Solution (ORS) is recommended by burn experts and professional burn societies when resources and access to intravenous fluid resuscitation are not available. Studies have previously demonstrated the efficacy and safety of enteral-based resuscitation in controlled, high-resource settings, however, there have not been real-world effectiveness trials in resource-constrained settings. Therefore, the investigators seek to ultimately address the problem of pre-hospital and pre-burn center admission resuscitation by studying the effectiveness of enteral resuscitation with Oral Rehydration Solution (ORS) in preventing burn shock. A recent feasibility and pilot study(n=30) of this Enteral-based implementation bundle (EResus) i.e., training resources, protocol, and toolkit were conducted. The pilot study allowed for protocol development and testing, established the feasibility, provided key insights into implementation and helped develop infrastructure and study standard operating procedures at the study site. With the current study, the investigators aim to expand the trial to a full effectiveness-implementation trial, which will allow to further hone the EResus protocol and bundle, generate more effective implementation strategies, and obtain a clearer understanding of efficacy and frequency of specific outcomes.

This study examines enteral-based resuscitation (i.e. enteral with/without IV Fluids) versus enhanced standard of care IV Fluids for the treatment of major burn injuries. The intervention portion of the study will entail randomization of patients presenting with acute burn injuries of 15-40% total body surface area (TBSA) to an enteral-based resuscitation versus the standard of care IV fluid resuscitation. The intervention will continue through the acute resuscitation period.

The primary study variables will include measures of urine output, vital signs, planned and administered resuscitation volumes, and routes of resuscitation along with frequency, timing, and treatment of any gastrointestinal symptomology, and serious adverse events such as kidney injury and aspiration events

Further, there will be a qualitative component to the study with focus group discussions of the bedside healthcare providers (doctors and nurses) caring for the enrolled patients, in order to understand the challenges and facilitators of enteral resuscitation. In-depth interviews will be conducted with enrolled patients and their families to further understand the patient perception, experience and challenges and facilitators. Qualitative analysis will be done to understand the major themes of challenges and facilitators to enteral resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with moderate-sized burn injuries [15- 40% total body surface areas (TBSA)] to the Nepal Cleft and Burn Center within 24 hours of injury.
* All gender

Exclusion Criteria:

* Breastfeeding patients
* Patients with electrical burns, chemical burns, and suspected severe inhalation injuries.
* Patients in overt shock (defined as serum lactate >2.5, or hypotension and altered mental status).
* Pregnant patients
* Patients with oropharyngeal defects and/or previously known diagnoses leading to a high risk of aspiration, and/or precluding safe nasal-enteric access will be excluded.
* Patients and/or family members who are unable to understand and provide informed consent for data abstraction or the interview will be excluded.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of enteral-based resuscitation | 2 years
  Measure the frequency of successful resuscitation for both enteral-based and IV fluid resuscitation protocols by measuring frequency of achieving goal average urine output of at least 0.5 mL/kg/hr per the resuscitation protocol for the overall 24 hour time period for each patient in the IV-fluid based and enteral-based resuscitation protocol arms as demonstrated on the Documentation Chart. This value will be calculated by taking the sum total of urine produced in milliliters during the resuscitation period (mL), divided by the patient's measured weight on admission in kilograms (kg), and further divided by the length of the resuscitation in hours (hr).
  The overall urine output in the resuscitation will be calculated for each patient. Based on the urine output and whether it achieved goal (0.5 mL/kg/hr) or not, each will be designated as "successful" or "unsuccessful". For each intervention arm, the proportion of patients with "successful" resuscitation will be calculated.
Challenges and facilitators to enteral-based resuscitation and IV fluid resuscitation protocols | 2 years
  These are qualitative metrics of the challenges and facilitators of adherance to the IV fluid and enteral-based resuscitation protocols as described by the clinical bedside providers. These will be obtained from focus group interviews with the bedside burn care providers at the study site. The focus group interviews will occur prior to patient enrollment, halfway through patient enrollment and after the conclusion of patient enrollment. The focus group interviews will be audiorecorded, and then will undergo transcription and translated as needed for qualitative thematic analysis.
  A codebook will be developed and thematic analysis conducted to understand the qualitative frequency and relevancy of each cited "challenge" and "facilitator" for adhering to the resuscitation protocols. These qualitative measures will not be graded with a score, or on a scale.

SECONDARY OUTCOMES:
Frequency of protocol adherence for recommended fluid adjustments | 2 years
  Measured frequency of adherence to the recommend fluid adjustments for both enteral-based resuscitation and IV fluid resuscitation protocols by measuring completion rate of appropriate fluid rate adjustments made, as documented in the Documentation Chart for each patient.
  The Documentation Chart will be analyzed for correct ("appropriate") adjustment at each time check interval (every 2 hours for adults >18years,every 1 hour for Pediatric group <18 years) during the resuscitation period, as demonstrated by fluid adjustment documentation on the Documentation Chart. The assessment will be reported as the proportion of "'appropriate" fluid adjustments out of total fluid adjustments, for each patient in the IV fluid resuscitation arm and each patient in the Enteral-based resuscitation arm.
Frequency of protocol adherence for documentation | 2 years
  Measured frequency of adherence to both enteral-based resuscitation and IV fluid resuscitation protocols by measuring completeness of documentation based on the proportion of rows filled out on the Documentation Chart during the acute resuscitation time period. This assessment will be reported as a proportion (percentage), and with a range from 0-100 percent, for each patient in the IV fluid resuscitation intervention arm and each patient in the Enteral-based resuscitation intervention arm.
Frequency of protocol adherence for laboratory assessments | 2 years
  Measured frequency of adherence to both enteral-based resuscitation and IV fluid resuscitation protocols by measuring completion rate of the recommended 8-hourly laboratory assessments as documented on the laboratory section of the Documentation Chart. The completeness will be measured based on the proportion of rows filled out in the laboratory section of the Documentation Chart during the acute resuscitation time period. This assessment will be reported as a proportion (percentage), and with a range from 0-100 percent, for each patient in the IV fluid resuscitation intervention arm and each patient in the enteral-based resuscitation intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran K Nakarmi, MBBS,MCh, Principal Investigator — Nepal Cleft and Burn Center,Kirtipur Hospital
Locations (1):
- Nepal Cleft and Burn Center, Kirtipur Hospital, Ki̇̄rtipur, Bagmati, Nepal